CLINICAL TRIAL: NCT00329238
Title: A Phase III, Randomised, Multicenter, Double-blind, Parallel-group, Active Controlled Study to Evaluate the Efficacy and Safety of Oral Dabigatran Etexilate (150 mg Bid) Compared to Warfarin (INR 2.0-3.0) for the Secondary Prevention of Venous Thromboembolism.
Brief Title: Secondary Prevention of Venous Thrombo Embolism (VTE).
Acronym: RE-MEDY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.47; 2005-002536-94 (EudraCT Number: EudraCT)
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Results first posted 2011-09-14 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2013-12

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Dabigatran; Warfarin

ARMS (2):
- Dabigatran (Experimental): Patient to receive 1 capsule containing dabigatran 150 mg twice daily plus placebo tablets for warfarin as decided by sham INR measurements
  Interventions: Drug: Dabigatran
- Warfarin (INR of 2.0-3.0) (Active Comparator): Patient to receive warfarin tablets to target INR 2.0-3.0 plus placebo capsules for dabigatran twice daily
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran — Dabigatran 150 mg BID (twice daily)
  Arms: Dabigatran
Drug: Warfarin — Warfarin dosed individually to maintain INR 2.0-3.0
  Arms: Warfarin (INR of 2.0-3.0)

SUMMARY:
The general aim of this study is to determine the comparative safety and efficacy of dabigatran etexilate administered orally and warfarin (International Normalized Ratio (INR) of 2.0-3.0) for the long-term treatment and secondary prevention of symptomatic venous thromboembolism in patients who have been successfully treated with standard doses of an approved anticoagulant for three to twelve months for confirmed acute symptomatic Venous Thrombo-embolism.

ELIGIBILITY:
Inclusion criteria:

Inclusion_Criteria

* Acute symptomatic deep vein thrombosis (DVT)
* Pulmonary embolism (PE) 3-12 months prior to screening, which has been documented by objective testing

Exclusion criteria:

Exclusion_Criteria

* Symptomatic DVT or PE at screening Interruption of anticoagulant therapy for 2 or more weeks during the 3-12 months of treatment for the prior VTE.
* Patients who in the investigators judgement are perceived as having an excessive risk of bleeding Elevated Aspartate aminotransferase (AST) or Alanine tranminase (ALT) > 2x ULN
* Severe renal impairment (estimated creatinine clearance <= 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2867 (Actual)
Dates: Start 2006-05; Primary Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (275):
- United States (18):
  - 1160.47.01035 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1160.47.01056 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 1160.47.01044 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.47.01019 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 1160.47.01008 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1160.47.01014 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.47.01018 Boehringer Ingelheim Investigational Site, Roxbury Crossing, Massachusetts
  - 1160.47.01023 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1160.47.01009 Boehringer Ingelheim Investigational Site, Saint Louis Park, Minnesota
  - 1160.47.01031 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 1160.47.01036 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1160.47.01027 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 1160.47.01039 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1160.47.01030 Boehringer Ingelheim Investigational Site, Grand Forks, North Dakota
  - 1160.47.01013 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1160.47.01052 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1160.47.01055 Boehringer Ingelheim Investigational Site, Summerville, South Carolina
  - 1160.47.01017 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Argentina (14):
  - 1160.47.54017 Boehringer Ingelheim Investigational Site, Adrogué
  - 1160.47.54015 Boehringer Ingelheim Investigational Site, Bahía Blanca
  - 1160.47.54001 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.47.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.47.54005 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.47.54006 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.47.54007 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.47.54010 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.47.54016 Boehringer Ingelheim Investigational Site, La Plata
  - 1160.47.54014 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1160.47.54013 Boehringer Ingelheim Investigational Site, Quilmes
  - 1160.47.54011 Boehringer Ingelheim Investigational Site, Rosario
  - 1160.47.54018 Boehringer Ingelheim Investigational Site, Salta
  - 1160.47.54012 Boehringer Ingelheim Investigational Site, Santa Fe
- Australia (6):
  - 1160.47.61002 Princess Alexandra Hospital, Wooloongabba, Queensland
  - 1160.47.61004 Boehringer Ingelheim Investigational Site, Bedford Park, South Australia
  - 1160.47.61003 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1160.47.61001 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1160.47.61006 Boehringer Ingelheim Investigational Site, Windsor, Victoria
  - 1160.47.61005 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Austria (4):
  - 1160.47.43001 Boehringer Ingelheim Investigational Site, Graz
  - 1160.47.43003 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1160.47.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.47.43004 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (4):
  - 1160.47.32001 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.47.32002 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.47.32005 Boehringer Ingelheim Investigational Site, Leuven
  - 1160.47.32004 Boehringer Ingelheim Investigational Site, Liège
- Brazil (8):
  - 1160.47.55010 Boehringer Ingelheim Investigational Site, Brasília
  - 1160.47.55007 Boehringer Ingelheim Investigational Site, Campinas - SP
  - 1160.47.55014 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.47.55017 Boehringer Ingelheim Investigational Site, Juvene - Paraná -
  - 1160.47.55012 Boehringer Ingelheim Investigational Site, pTO aLEGRE
  - 1160.47.55016 Boehringer Ingelheim Investigational Site, Rio de Janeiro - RJ
  - 1160.47.55018 Boehringer Ingelheim Investigational Site, São Bernardo do Campo
  - 1160.47.55005 Boehringer Ingelheim Investigational Site, São José do Rio Preto
- Bulgaria (8):
  - 1160.47.35910 Boehringer Ingelheim Investigational Site, Plovdiv
  - 1160.47.35908 Boehringer Ingelheim Investigational Site, Rousse
  - 1160.47.35901 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.47.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.47.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.47.35906 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.47.35907 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.47.35905 Boehringer Ingelheim Investigational Site, Varna
- Canada (15):
  - 1160.47.02006 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.47.02013 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.47.02021 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1160.47.02004 Boehringer Ingelheim Investigational Site, Saint Johns, New Brunswick
  - 1160.47.02001 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1160.47.02002 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.47.02005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.47.02010 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.47.02022 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.47.02015 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1160.47.02019 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.47.02008 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.47.02009 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.47.02014 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.47.02017 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- China (15):
  - 1160.47.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.47.86015 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.47.86014 Boehringer Ingelheim Investigational Site, Chengdu
  - 1160.47.86012 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1160.47.86009 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1160.47.86010 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1160.47.86013 Boehringer Ingelheim Investigational Site, Nanjing
  - 1160.47.86002 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.47.86003 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.47.86004 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.47.86005 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.47.86006 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.47.86007 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.47.86016 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.47.86011 Boehringer Ingelheim Investigational Site, Shijiazhuang
- Czechia (10):
  - 1160.47.42001 Boehringer Ingelheim Investigational Site, Brno
  - 1160.47.42002 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1160.47.42011 Boehringer Ingelheim Investigational Site, Hranice
  - 1160.47.42012 Boehringer Ingelheim Investigational Site, Liberec
  - 1160.47.42015 Boehringer Ingelheim Investigational Site, Nový Jičín
  - 1160.47.42005 Boehringer Ingelheim Investigational Site, Ostrava-Vitkovice
  - 1160.47.42004 Boehringer Ingelheim Investigational Site, Prague
  - 1160.47.42014 Boehringer Ingelheim Investigational Site, Tábor
  - 1160.47.42010 Boehringer Ingelheim Investigational Site, Ústí nad Labem
  - 1160.47.42007 Boehringer Ingelheim Investigational Site, Zlín
- Denmark (6):
  - 1160.47.45008 Boehringer Ingelheim Investigational Site, Esbjerg
  - 1160.47.45009 Boehringer Ingelheim Investigational Site, Holbæk
  - 1160.47.45002 Boehringer Ingelheim Investigational Site, Kolding
  - 1160.47.45004 Boehringer Ingelheim Investigational Site, København NV
  - 1160.47.45007 Boehringer Ingelheim Investigational Site, København S
  - 1160.47.45006 Boehringer Ingelheim Investigational Site, Slagelse
- Finland (5):
  - 1160.47.35804 Boehringer Ingelheim Investigational Site, Espoo
  - 1160.47.35801 Boehringer Ingelheim Investigational Site, Helsinki
  - 1160.47.35802 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1160.47.35805 Boehringer Ingelheim Investigational Site, Kuopio
  - 1160.47.35803 Boehringer Ingelheim Investigational Site, Tampere
- France (14):
  - 1160.47.3301A Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3301B Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3301C Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3301D Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3301E Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3301F Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3301H Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3301I Boehringer Ingelheim Investigational Site, Brest
  - 1160.47.3302A Boehringer Ingelheim Investigational Site, Lorient
  - 1160.47.3303A Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.47.3303B Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.47.3303C Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.47.3303D Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.47.3308A Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (8):
  - 1160.47.49003 Boehringer Ingelheim Investigational Site, Cologne
  - 1160.47.49017 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.47.49018 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.47.49005 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.47.49006 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.47.49007 Boehringer Ingelheim Investigational Site, München
  - 1160.47.49008 Boehringer Ingelheim Investigational Site, München
  - 1160.47.49009 Boehringer Ingelheim Investigational Site, Püttlingen
- Greece (4):
  - 1160.47.30001 Boehringer Ingelheim Investigational Site, Athens
  - 1160.47.30006 Boehringer Ingelheim Investigational Site, Athens
  - 1160.47.30007 Boehringer Ingelheim Investigational Site, Athens
  - 1160.47.30009 Boehringer Ingelheim Investigational Site, Athens
- Hungary (9):
  - 1160.47.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.47.36006 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.47.36007 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.47.36002 Boehringer Ingelheim Investigational Site, Debrecen
  - 1160.47.36012 Boehringer Ingelheim Investigational Site, Gyula
  - 1160.47.36004 Boehringer Ingelheim Investigational Site, Miskolc
  - 1160.47.36003 Boehringer Ingelheim Investigational Site, Pécs
  - 1160.47.36010 Boehringer Ingelheim Investigational Site, Székesfehérvár
  - 1160.47.36011 Boehringer Ingelheim Investigational Site, Szombathely
- India (15):
  - 1160.47.91002 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1160.47.91011 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.47.91015 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.47.91012 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.47.91017 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.47.91009 Boehringer Ingelheim Investigational Site, Madurai
  - 1160.47.91007 Boehringer Ingelheim Investigational Site, Mysore
  - 1160.47.91003 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.47.91006 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.47.91010 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.47.91001 Boehringer Ingelheim Investigational Site, Pune
  - 1160.47.91005 Boehringer Ingelheim Investigational Site, Pune
  - 1160.47.91008 Boehringer Ingelheim Investigational Site, Pune
  - 1160.47.91014 Boehringer Ingelheim Investigational Site, Trivandrum
  - 1160.47.91004 Boehringer Ingelheim Investigational Site, Vadodara
- Israel (10):
  - 1160.47.97202 Boehringer Ingelheim Investigational Site, Afula
  - 1160.47.97207 Boehringer Ingelheim Investigational Site, Ashkelon
  - 1160.47.97211 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.47.97203 Boehringer Ingelheim Investigational Site, Holon
  - 1160.47.97205 Boehringer Ingelheim Investigational Site, Kfar Saba
  - 1160.47.97206 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1160.47.97208 Boehringer Ingelheim Investigational Site, Rehovot
  - 1160.47.97210 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.47.97204 Boehringer Ingelheim Investigational Site, Tel Litwinsky
  - 1160.47.97201 Boehringer Ingelheim Investigational Site, Ẕerifin
- Italy (7):
  - 1160.47.39003 Boehringer Ingelheim Investigational Site, Bologna
  - 1160.47.39004 Boehringer Ingelheim Investigational Site, Cremona
  - 1160.47.39006 Boehringer Ingelheim Investigational Site, Genova
  - 1160.47.39008 Boehringer Ingelheim Investigational Site, Milan
  - 1160.47.39007 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 1160.47.39009 Boehringer Ingelheim Investigational Site, Udine
  - 1160.47.39005 Boehringer Ingelheim Investigational Site, Vittorio Veneto
- Mexico (5):
  - 1160.47.52036 Boehringer Ingelheim Investigational Site, Chihuahua City
  - 1160.47.52039 Boehringer Ingelheim Investigational Site, Culiacán
  - 1160.47.52030 Boehringer Ingelheim Investigational Site, Guadalajara, Jal.
  - 1160.47.52027 Boehringer Ingelheim Investigational Site, Monterrey
  - 1160.47.52034 Boehringer Ingelheim Investigational Site, San Luis Potosí City
- Netherlands (8):
  - 1160.47.31010 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1160.47.31001 Boehringer Ingelheim Investigational Site, Amersfoort
  - 1160.47.31006 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.47.31007 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.47.31014 Boehringer Ingelheim Investigational Site, Heerlen
  - 1160.47.31005 Boehringer Ingelheim Investigational Site, Maastricht
  - 1160.47.31004 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1160.47.31009 Boehringer Ingelheim Investigational Site, Rotterdam
- New Zealand (4):
  - 1160.47.64004 Boehringer Ingelheim Investigational Site, Christchurch
  - 1160.47.64003 Boehringer Ingelheim Investigational Site, Grafton
  - 1160.47.64002 Boehringer Ingelheim Investigational Site, Otahuhu
  - 1160.47.64001 Boehringer Ingelheim Investigational Site, Takapuna Auckland 9
- Norway (4):
  - 1160.47.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.47.47004 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.47.47003 Boehringer Ingelheim Investigational Site, Rud
  - 1160.47.47005 Boehringer Ingelheim Investigational Site, Trondheim
- Poland (5):
  - 1160.47.48004 Boehringer Ingelheim Investigational Site, Kielce
  - 1160.47.48005 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.47.48007 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.47.48003 Boehringer Ingelheim Investigational Site, Poznan
  - 1160.47.48006 Boehringer Ingelheim Investigational Site, Warsaw
- Portugal (6):
  - 1160.47.35104 Boehringer Ingelheim Investigational Site, Almada
  - 1160.47.35109 Boehringer Ingelheim Investigational Site, Coimbra
  - 1160.47.35107 Boehringer Ingelheim Investigational Site, Covilha
  - 1160.47.35101 Boehringer Ingelheim Investigational Site, Lisbon
  - 1160.47.35102 Boehringer Ingelheim Investigational Site, Lisbon
  - 1160.47.35105 Boehringer Ingelheim Investigational Site, Lisbon
- Russia (20):
  - 1160.47.07022 Boehringer Ingelheim Investigational Site, Belgorod
  - 1160.47.07011 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1160.47.07021 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1160.47.07016 Boehringer Ingelheim Investigational Site, Krasnodar
  - 1160.47.07004 Boehringer Ingelheim Investigational Site, Kursk
  - 1160.47.07010 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1160.47.07020 Boehringer Ingelheim Investigational Site, Omsk
  - 1160.47.07018 Boehringer Ingelheim Investigational Site, Pskov
  - 1160.47.07009 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.47.07023 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.47.07024 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.47.07025 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.47.07001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.47.07002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.47.07017 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.47.07019 Boehringer Ingelheim Investigational Site, Tyumen
  - 1160.47.07014 Boehringer Ingelheim Investigational Site, Ufa
  - 1160.47.07005 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.47.07006 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.47.07007 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Slovakia (5):
  - 1160.47.42107 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1160.47.42106 Boehringer Ingelheim Investigational Site, Lučenec
  - 1160.47.42102 Boehringer Ingelheim Investigational Site, Nitra
  - 1160.47.42103 Boehringer Ingelheim Investigational Site, Nové Zámky
  - 1160.47.42104 Boehringer Ingelheim Investigational Site, Žilina
- South Africa (6):
  - 1160.47.27001 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.47.27002 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.47.27006 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.47.27007, Pretoria
  - 1160.47.27003 Boehringer Ingelheim Investigational Site, Randburg
  - 1160.47.27005 Boehringer Ingelheim Investigational Site, Roodepoort
- Spain (9):
  - 1160.47.34006 Boehringer Ingelheim Investigational Site, Alicante
  - 1160.47.34012 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 1160.47.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.47.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.47.34007 Boehringer Ingelheim Investigational Site, Cartagena. Murcia
  - 1160.47.34003 Boehringer Ingelheim Investigational Site, Cuenca
  - 1160.47.34009 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.47.34004 Boehringer Ingelheim Investigational Site, Santander
  - 1160.47.34011 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (7):
  - 1160.47.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.47.46006 Boehringer Ingelheim Investigational Site, Jönköping
  - 1160.47.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.47.46007 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.47.46008 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.47.46005 Boehringer Ingelheim Investigational Site, Sundsvall
  - 1160.47.46003 Boehringer Ingelheim Investigational Site, Uppsala
- Turkey (Türkiye) (7):
  - 1160.47.90003 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.47.90004 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.47.90005 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.47.90001 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.47.90002 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.47.90007 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.47.90006 Boehringer Ingelheim Investigational Site, Izmir
- Ukraine (4):
  - 1160.47.38002 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1160.47.38006 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.47.38005 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1160.47.38003 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (5):
  - 1160.47.44005 Boehringer Ingelheim Investigational Site, Headington, Oxford
  - 1160.47.44009 Boehringer Ingelheim Investigational Site, London
  - 1160.47.44011 Boehringer Ingelheim Investigational Site, London
  - 1160.47.44006 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1160.47.44012 Boehringer Ingelheim Investigational Site, Sheffield

REFERENCES:
- [Derived] Goldhaber SZ, Eriksson H, Kakkar A, Schellong S, Feuring M, Fraessdorf M, Kreuzer J, Schueler E, Schulman S. Efficacy of dabigatran versus warfarin in patients with acute venous thromboembolism in the presence of thrombophilia: Findings from RE-COVER(R), RE-COVER II, and RE-MEDY. Vasc Med. 2016 Dec;21(6):506-514. doi: 10.1177/1358863X16668588. Epub 2016 Nov 1. PMID 27807306
- [Derived] Majeed A, Hwang HG, Connolly SJ, Eikelboom JW, Ezekowitz MD, Wallentin L, Brueckmann M, Fraessdorf M, Yusuf S, Schulman S. Management and outcomes of major bleeding during treatment with dabigatran or warfarin. Circulation. 2013 Nov 19;128(21):2325-32. doi: 10.1161/CIRCULATIONAHA.113.002332. Epub 2013 Sep 30. PMID 24081972
- [Derived] Schulman S, Kearon C, Kakkar AK, Schellong S, Eriksson H, Baanstra D, Kvamme AM, Friedman J, Mismetti P, Goldhaber SZ; RE-MEDY Trial Investigators; RE-SONATE Trial Investigators. Extended use of dabigatran, warfarin, or placebo in venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):709-18. doi: 10.1056/NEJMoa1113697. PMID 23425163

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran: 150 mg twice daily, total daily dose 300 mg
- Warfarin: Target International Normalized Ratio (INR) of 2.0 to 3.0
Period: Overall Study
Arm/Group | Dabigatran | Warfarin
Started | 1430 (2866 were randomized. A total of ten did not receive treatment resulting in 2856 starting study.) | 1426 (2866 were randomized. A total of ten did not receive treatment resulting in 2856 starting study.)
Completed | 1154 | 1145
Not Completed | 276 | 281
Not completed — Adverse Event | 147 | 129
Not completed — Protocol Violation | 23 | 34
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 64 | 58
Not completed — Other reason (not specified) | 40 | 54

BASELINE CHARACTERISTICS:
Population: The FAS consisted of all randomised patients who were documented to have taken at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Warfarin | Total
Number analyzed (Participants) | 1430 | 1426 | 2856
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.38 (14.99) | 53.90 (15.34) | 54.64 (15.18)
Age, Customized [Number; unit: participants]
  >=18 to <40 years | 237 | 269 | 506
  >=40 to <50 years | 250 | 291 | 541
  >=50 to <65 years | 500 | 459 | 959
  >=65 to <75 years | 303 | 288 | 591
  >= 75 years | 140 | 119 | 259
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 559 | 555 | 1114
  Male | 871 | 871 | 1742
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic/Latino | 1325 | 1317 | 2642
  Hispanic/Latino | 105 | 109 | 214
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1288 | 1284 | 2572
  Black | 29 | 28 | 57
  Asian | 113 | 114 | 227
Height [Mean (Standard Deviation); unit: cm] — N = 1429, 1424, 2853
  cm | 171.55 (9.73) | 171.95 (10.08) | 171.75 (9.90)
Weight [Mean (Standard Deviation); unit: kg] — N = 1429, 1422, 2851
  kg | 86.09 (19.26) | 85.95 (18.87) | 86.02 (19.06)
Weight category [Number; unit: Participants]
  < 50 kg | 10 | 5 | 15
  >= 50 to < 100 kg | 1120 | 1117 | 2237
  >= 100 kg | 299 | 300 | 599
  Missing | 1 | 4 | 5
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/square meter] — N = 1428, 1422, 2850
  kg/square meter | 29.15 (5.65) | 29.01 (5.75) | 29.08 (5.70)
Body Mass Index (BMI) category [Number; unit: Participants]
  <25 kg/square meter | 315 | 334 | 649
  >=25 to <30 kg/square meter | 571 | 584 | 1155
  >=30 to <35 kg/square meter | 356 | 330 | 686
  >= 35 kg/square meter | 186 | 174 | 360
  Missing | 2 | 4 | 6
Smoking history [Number; unit: Participants]
  Non-smoker | 814 | 829 | 1643
  Ex-smoker | 393 | 366 | 759
  Current smoker | 223 | 231 | 454
Serum creatinine clearance [Mean (Standard Deviation); unit: mL/min] — N = 1418, 1410, 2828
  mL/min | 104.2 (38.6) | 106.6 (37.9) | 105.4 (38.3)
Serum creatinine clearance category [Number; unit: Participants]
  >=0 to <30 mL/min | 0 | 4 | 4
  >=30 to <50 mL/min | 59 | 45 | 104
  >=50 to <80 mL/min | 328 | 289 | 617
  >= 80 mL/min | 1031 | 1072 | 2103
  Missing | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Composite of Recurrent VTE or VTE Death at 36 Months
Description: Endpoint is a composite of recurrent Venous Thromboembolic Event (VTE) and death related to VTE. VTE was defined as the composite of symptomatic Deep Vein Thrombosis (DVT) of the leg and Pulmonary embolism (PE). All recurrent VTEs required objective verification by definitive diagnostic evaluation. In case of death, autopsy was an additional way to confirm VTE.
Time Frame: 36 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 26 | 18
  Number of participants with no event | 1404 | 1408
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Non-Inferiority or Equivalence — Comparisons between treatment groups were performed using a Cox regression analysis with treatment and baseline stratification factor in the model; p = 0.0137, Regression, Cox — p-value for non-inferiority. The non-inferiority margin for the hazard ratio was chosen to be 2.85; HR within cohort estimated by Cox regr. with treatment and baseline stratific. factor. Overall HR calc. by pooling with inverse variance weighting; Hazard Ratio (HR) = 1.44, 95% CI [0.78 to 2.64] — HR for time to first recurrent VTE or VTE death
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; p = 0.2424, Regression, Cox — p-value for superiority. If non-inferiority could be established for HR and for the risk difference, the upper bound of the 95% CI for the hazard ratio was then compared with 1 to evaluate the superiority claim of dabigatran over warfarin

2. Primary Outcome: Composite of Recurrent VTE or VTE Death at 18 Months
Description: as for outcome 1
Time Frame: 18 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 22 | 17
  Number of participants with no event | 1408 | 1409
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Cox — p-value for non-inferiority. The non-inferiority margin for the risk difference was chosen to be 2.80; Risk difference for time to first recurrent VTE/VTE death is calculated based on weighted KM estimates across the cohorts via meta-analysis approach; Risk Difference (RD) = 0.38, 95% CI [-0.50 to 1.25]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; p = 0.4013, Kaplan-Meier — p-value for superiority. If non-inferiority could be established for HR and for the risk difference, the upper bound of the 95% CI for the risk difference was then compared with 0 to evaluate the superiority claim of dabigatran over warfarin

3. Secondary Outcome: Composite of Recurrent VTE or All Cause Death at 36 Months
Description: Endpoint is a composite of recurrent Venous Thromboembolic Event (VTE) and all cause death. VTE was defined as the composite of symptomatic Deep Vein Thrombosis (DVT) of the leg and Pulmonary embolism (PE). All recurrent VTEs required objective verification by definitive diagnostic evaluation.
Time Frame: 36 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 42 | 36
  Number of participants with no event | 1388 | 1390
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Test type: Superiority or Other; p = 0.4732, Regression, Cox; Hazard ratio estimated using the Cox regression with treatment, cohort, baseline stratification factors and their interaction; Hazard Ratio (HR) = 1.18, 95% CI [0.75 to 1.84] — HR for time to first centrally adjudicated recurrent VTE or all cause death

4. Secondary Outcome: Composite of Recurrent VTE or All Cause Death at 18 Months
Description: as for outcome 3
Time Frame: 18 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 36 | 32
  Number of participants with no event | 1394 | 1394
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.8876, Kaplan-Meier; Risk difference for the time to first centrally adjudicated recurrent VTE or all cause death at month 18; Risk Difference (RD) = 0.09, 95% CI [-1.11 to 1.28]

5. Secondary Outcome: Deep Vein Thrombosis (DVT) at 36 Months
Description: Symptomatic Deep vein thrombosis (DVT). All DVT events required objective verification through definitive diagnostic evaluation.
Time Frame: 36 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 17 | 13
  Number of participants with no event | 1413 | 1413
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.4548, Regression, Cox; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.32, 95% CI [0.64 to 2.71] — HR for time to first centrally adjudicated recurrent symptomatic DVT

6. Secondary Outcome: DVT at 18 Months
Description: as for outcome 5
Time Frame: 18 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 15 | 12
  Number of participants with no event | 1415 | 1414
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.6563, Kaplan-Meier; Risk difference for the time to first centrally adjudicated recurrent symptomatic DVT at Month 18; Risk Difference (RD) = 0.19, 95% CI [-0.63 to 1.00]

7. Secondary Outcome: Symptomatic Pulmonary Embolism (PE) at 36 Months
Description: Symptomatic pulmonary embolism (PE) at 36 Months (fatal or non-fatal). All suspected PEs required confirmation by one of the following: ventilation-perfusion (V-Q) lung scan, pulmonary angiography, or spiral (helical) Computed tomography.
Time Frame: 36 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 10 | 5
  Number of participants with no event | 1420 | 1421
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.1925, Regression, Cox; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 2.04, 95% CI [0.70 to 5.98] — Hazard ratio for time to first centrally adjudicated recurrent symptomatic PE

8. Secondary Outcome: Symptomatic Pulmonary Embolism (PE) at 18 Months
Description: Symptomatic pulmonary embolism (PE) at 18 Months (fatal or non-fatal). All suspected PEs required confirmation by one of the following: ventilation-perfusion (V-Q) lung scan, pulmonary angiography, or spiral (helical) Computed tomography.
Time Frame: 18 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 8 | 5
  Number of participants with no event | 1422 | 1421
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.3723, Kaplan-Meier; Risk Difference (RD) = 0.26, 95% CI [-0.32 to 0.84] — Risk difference for the time to first centrally adjudicated recurrent symptomatic PE at Month 18

9. Secondary Outcome: Deaths Related to VTE at 36 Months
Description: Deaths related to VTE (i.e. fatal PE) at 36 Months. Deaths related to VTE (i.e. fatal PE) at 18 Months. All deaths were centrally adjudicated by the Independent Central Adjudication Committee for VTE and death in a treatment-blinded way.
Time Frame: 36 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 1 | 1
  Number of participants with no event | 1429 | 1425
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.9921, Regression, Cox; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI [0.06 to 16.22] — Hazard ratio for time to deaths related to VTE

10. Secondary Outcome: Deaths Related to VTE at 18 Months
Description: Deaths related to VTE (i.e. fatal PE) at 18 Months. All deaths were centrally adjudicated by the Independent Central Adjudication Committee for VTE and death in a treatment-blinded way.
Time Frame: 18 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 1 | 1
  Number of participants with no event | 1429 | 1425
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.9204, Kaplan-Meier; Risk difference for the time to deaths related to VTE at Month 18; Risk Difference (RD) = 0.01, 95% CI [-0.20 to 0.23]

11. Secondary Outcome: Deaths of All Causes at 36 Months
Description: Deaths of all causes at 36 Months. All components of the primary efficacy endpoint and all deaths were centrally adjudicated by the Independent Central Adjudication Committee for VTE and death without knowledge of any individual treatment assignments.
Time Frame: 36 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 17 | 19
  Number of participants with no event | 1413 | 1407
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.7405, Regression, Cox; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI [0.47 to 1.72] — Hazard ratio for time to all deaths

12. Secondary Outcome: Deaths of All Causes at 18 Months
Description: Deaths of all causes at 18 Months. All components of the primary efficacy endpoint and all deaths were centrally adjudicated by the Independent Central Adjudication Committee for VTE and death without knowledge of any individual treatment assignments.
Time Frame: 18 months
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
Participants
  Number of participants with event | 15 | 16
  Number of participants with no event | 1415 | 1410
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Dabigatran versus Warfarin; Test type: Superiority or Other; p = 0.9622, Kaplan-Meier; Risk difference for the time to all deaths at Month 18; Risk Difference (RD) = -0.02, 95% CI [-0.89 to 0.84]

13. Secondary Outcome: Number of Participants With Bleeding Events
Description: MBE (major bleeding event) if it fulfilled at least one of the following criteria
  * Fatal bleeding
  * Symptomatic bleeding in a critical area or organ.
  * Bleeding causing a fall in haemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of 2 or more units of whole blood or red cells.
  Minor bleeding event was any bleeding that did not fulfil any of the criteria for MBEs
  CRBE (clinically relevant bleeding event) if it is a minor bleeding events which fulfilled at least one of the following criteria
  * Spontaneous skin haematoma ≥25 cm2
  * Spontaneous nose bleed >5 min duration
  * Macroscopic haematuria, either spontaneous or, if associated with an intervention, lasting >24 h
  * Spontaneous rectal bleeding
  * Gingival bleeding >5 min
  * Bleeding leading to hospitalisation or requiring surgical treatment
  * Bleeding leading to a transfusion of <2 units of whole blood or red cells
  * Any other bleeding event considered clinically relevant by the investigator
Time Frame: first intake of study drug until 6 days following last intake of study drug
Population: FAS as treated
Measure: Number; unit: participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1426
participants
  patients with MBE | 13 | 25
  patients with MBE and /or CRBE | 80 | 145
  patients with any bleeding event | 277 | 373
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Hazard ratio estimated using the Cox regression with treatment, cohort, baseline stratification factors (including active cancer at baseline and symptomatic PE as qualifying event) and their interaction; Test type: Superiority or Other; p = 0.0577, Regression, Cox; Hazard Ratio (HR) = 0.52, 95% CI [0.27 to 1.02] — This is the analysis of the time to the first MBE
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.61 to 0.83] — This is the analysis of the time to the first occurrence of any bleeding event

14. Secondary Outcome: Laboratory Analysis
Description: Patients with LFT (liver function tests) increases of possible clinical significance during treatment. Increases of possible clinical significance were defined as: ≥3 x ULN (AST, ALT), ≥2 x ULN (AP), and ≥2 mg/dL (total bilirubin). Only patients with a baseline value which was not of possible clinical significance (or without any baseline value) could have a PCSA (Possible clinically significant abnormality).
Time Frame: 18 months + 30 days follow up
Population: FAS as treated
Measure: Number; unit: participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1411 | 1402
participants
  ALT increase | 26 | 30
  AST increase | 23 | 23
  Alkaline phosphatase | 9 | 14
  Total bilirubin | 9 | 8

15. Secondary Outcome: Number of Participants With Definite Acute Coronary Syndrome (ACS)
Description: All suspected ACS occurring during the trial were to be recorded on the CRF and were to be centrally adjudicated by an independent ACS/AC in a treatment-blinded manner.
Time Frame: day of first study drug intake until last day of study drug intake; from the day after last intake of study drug until trial termination
Population: FAS as treated
Measure: Number; unit: participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 1430 | 1415
participants
  During intake of study drug, N=1430 , N=1415 | 12 | 2
  After stopping study drug, N=1426, N=1400 | 1 | 5

ADVERSE EVENTS:
Time Frame: 18-month treatment period
Description: 30-day follow-up period subsequent to the completion of treatment
Arm/Group | Dabigatran | Warfarin | Post Dabigatran | Post Warfarin
Serious Adverse Events (participants affected / at risk) | 227/1430 | 224/1426 | 33/1395 | 41/1384
Other Adverse Events (participants affected / at risk) | 409/1430 | 415/1426 | 34/1395 | 32/1384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (N=1430) | Warfarin (N=1426) | Post Dabigatran (N=1395) | Post Warfarin (N=1384)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac asthma (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 3 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 3 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 6 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Metabolic myopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Retinal vascular thrombosis (Eye disorders) | 0 | 1 | 0 | 0
Trichiasis (Eye disorders) | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 2 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 8 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecal vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal strangulation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 2 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 4 | 1 | 0 | 0
Chest pain (General disorders) | 4 | 9 | 0 | 2
Death (General disorders) | 0 | 1 | 1 | 0
Device breakage (General disorders) | 0 | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 1 | 0
Diapedesis (General disorders) | 0 | 0 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0 | 0
Mass (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 4 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 3 | 1 | 1
Chronic hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 3 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 5 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 0 | 1
Endometritis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 3 | 3 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Gingival abscess (Infections and infestations) | 0 | 1 | 0 | 0
Gnathostomiasis (Infections and infestations) | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 2 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 5 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 1 | 0 | 0
Purulence (Infections and infestations) | 0 | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 1 | 0 | 3
Septic shock (Infections and infestations) | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Accidental drug intake by child (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 4 | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Arteriogram coronary normal (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0
Coagulation time prolonged (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 4 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to retroperitoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Omentum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid artery dissection (Nervous system disorders) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 2 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0
Diabetic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Facial neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 2 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 3 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 1
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 2 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 6 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 4 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Epididymal enlargement (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 3 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 3 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 2 | 2 | 1
Colostomy closure (Surgical and medical procedures) | 0 | 0 | 0 | 1
Femoral hernia repair (Surgical and medical procedures) | 0 | 1 | 0 | 0
Finger amputation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 2 | 0 | 0 | 0
Incisional hernia repair (Surgical and medical procedures) | 1 | 0 | 0 | 0
Joint arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 2 | 0 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aneurysm ruptured (Vascular disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 1 | 0 | 0
Arterial insufficiency (Vascular disorders) | 1 | 0 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0 | 1 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 10 | 6 | 1 | 2
Haematoma (Vascular disorders) | 0 | 3 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 2 | 0 | 1 | 0
Varicose ulceration (Vascular disorders) | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (N=1430) | Warfarin (N=1426) | Post Dabigatran (N=1395) | Post Warfarin (N=1384)
Diarrhoea (Gastrointestinal disorders) | 73 | 51 | 4 | 3
Oedema peripheral (General disorders) | 76 | 68 | 8 | 3
Influenza (Infections and infestations) | 75 | 67 | 2 | 11
Nasopharyngitis (Infections and infestations) | 112 | 127 | 5 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 109 | 110 | 9 | 6
Headache (Nervous system disorders) | 84 | 100 | 4 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 46 | 92 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.